CLINICAL TRIAL: NCT04022317
Title: A Randomised, Double-blind, Two-period Crossover, Euglycaemic Glucose Clamp Study in Healthy Volunteers to Demonstrate Pharmacokinetic and Pharmacodynamic Similarity of Biocon Insulin R and Humulin® R
Brief Title: Comparision of Pharmacokinetics(PK) and Pharmacodynamics(PD) of Biocon Insulin R and Humulin® R
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocon Limited (Industry)
Collaborators: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: EQR
Record Dates: First submitted 2019-06-29; First posted 2019-07-17 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Healthy Volunteer
Keywords: Recombinant Human Insulin R (rhi R)

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Biocon Insulin R (Experimental): 0.3 IU/kg Dose per administration, subcutaneous Route of administration
  Interventions: Biological: Biocon Insulin R
- Humulin® R (regular insulin human) (Active Comparator): 0.3 IU/kg Dose per administration, subcutaneous Route of administration
  Interventions: Biological: Humulin®R

INTERVENTIONS:
Biological: Biocon Insulin R — Biocon Insulin R is a short-acting human insulin, produced by recombinant deoxyribonucleic acid (rDNA) technology utilizing Pichia pastoris (yeast).
  Arms: Biocon Insulin R
Biological: Humulin®R — Humulin® R is a polypeptide hormone structurally identical to human insulin synthesised through recombinant deoxyribonucleic acid (rDNA) technology in a non-pathogenic laboratory strain of Escherichia coli bacteria.
  Arms: Humulin® R (regular insulin human)

SUMMARY:
Single-centre, randomised, double-blind, single dose, two-treatment, two-period, two sequence, crossover,12-hour euglycaemic glucose clamp trial in healthy subjects

DETAILED DESCRIPTION:
The present study is designed to demonstrate pharmacokinetic and pharmacodynamic equivalence of Biocon Insulin R with Humulin® R in healthy subjects.

The treatment consists of one single dose of the test or reference product, administered during each of the two study periods, separated by 5-7 days between each dosing.

The planned trial duration for each subject is about 12 to 36 days. Eligible subjects will undergo two 12-hour euglycaemic clamp examinations, one after administration of the test product and one after administration of the reference product in random order.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or post-menopausal female subject. Post-menopausal state is defined as no menses for 12 months without an alternative medical cause and confirmed by a follicle stimulating hormone (FSH) level in the post-menopausal range (>= 25.8 IU/L).
* Age between 18 and 55 years, both inclusive.
* Body Mass Index (BMI) between 18.5 and 29.0 kg/m^2, both inclusive.
* Fasting plasma glucose concentration <= 100 mg/dL.
* Considered generally healthy upon completion of medical history and screening safety assessments, as judged by the Investigator

Exclusion Criteria:

* Known or suspected hypersensitivity to Investigational Medicinal products (IMP(s)) or related products.
* Receipt of any medicinal product in clinical development within 30 days or five times its half-life (whichever is longer) before randomisation in this trial.
* Any history or presence of clinically relevant comorbidity, as judged by the investigator.
* Systolic blood pressure < 95 mmHg or >140 mmHg and/or diastolic blood pressure < 50 mm Hg or > 90 mmHg after resting for at least 5 minutes in supine position (excluding white-coat hypertension; therefore, a repeat test showing results within range will be acceptable).
* Pulse rate at rest outside the range of 50-90 beats per minute.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
PK endpoints:Area under the insulin concentration curve(AUCins).0-12h | 0-12 hours
  Area under the insulin concentration curve from 0 to 12 hours.
PD endpoints: Area under the glucose infusion rate curve(AUCGIR).0-12h | 0-12 hours
  Area under the glucose infusion rate curve
PK endpoints: Maximum observed insulin concentration(Cins.max) | 0-12 hours
  Maximum observed insulin concentration
PD endpoints:maximum glucose infusion rate(GIRmax) | 0-12 hours
  maximum glucose infusion rate

SECONDARY OUTCOMES:
PK endpoint- Area under the insulin concentration curve(AUCins).0-2h | 0 to 2 hours
  Area under the insulin concentration curve
PK endpoint- Area under the insulin concentration curve(AUCins).0-6h | 0 to 6 hours
  area under the insulin concentration curve
PK endpoint- Area under the insulin concentration curve(AUCins).6-12h | 6 to 12 hours
  area under the insulin concentration curve
PK endpoint- Area under the insulin concentration curve(AUCins).0-infinity | 0 hours to 24 hours
  area under the insulin concentration-time curve
PK endpoint- time to maximum concentration( tmax) | 0-12 hours
  time to maximum observed insulin concentration.
PK endpoint- time(t)50%-ins(early) | 0-12 hours
  time to half-maximum before Cins.max.
PK endpoint- time(t)50%-ins(late) | 0-12 hours
  time to half-maximum after Cins.max.
PK endpoint- terminal elimination half-life (t½) | 0-12 hours
  terminal elimination half-life calculated as t½=ln2/λz.
PK endpoint- terminal elimination rate constant (λz) | 0-12 hours
  terminal elimination rate constant of insulin.
PD endpoint: area under the glucose infusion rate curve(AUCGIR).0-2h | 0 to 2 hours
  area under the glucose infusion rate curve
PD endpoint: area under the glucose infusion rate curve(AUCGIR).0-6h | 0 to 6 hours
  area under the glucose infusion rate curve
PD endpoint: area under the glucose infusion rate curve(AUCGIR).6-12h | 6 to 12 hours
  area under the glucose infusion rate curve
PD endpoint: time to maximum glucose infusion rate (tGIR.max) | 0-12 hours
  time to maximum glucose infusion rate
PD endpoint: time to half-maximum glucose infusion rate before GIRmax (tGIR,50%-early | 0-12 hours
  time to half-maximum glucose infusion rate before GIRmax
PD endpoint:time to half-maximum glucose infusion rate after GIRmax (tGIR.50%-late) | 0-12 hours
  time to half-maximum glucose infusion rate after Maximum glucose infusion rate(GIRmax)
PD endpoint: Onset of action | 0-12 hours
  ime from trial product administration until blood glucose concentration has decreased at least 5 mg/dL from baseline, where baseline is defined as the mean of blood glucose levels from -6, -4, and -2 minutes before trial product administration as measured by ClampArt®((name of Clamp Devise)

OTHER OUTCOMES:
Safety endpoints: Number of subjects with Adverse Events, clinically significant changes in Physical examination, Vital signs. Local tolerability/ Injection site reactions | First dose to followup period (Total duration: 14 days approximate)
  Number of subjects with Adverse Events, clinically significant changes in Physical examination, Vital signs
  Local tolerability/ Injection site reactions
Safety endpoint: Number of subjects with clinically significant changes in Laboratory safety parameters, Electrocardiogram (ECG) | Screening to Follow-up period (Total duration: 35 days approximate)
  Number of subjects with clinically significant changes in Laboratory safety parameters.
  Number of subjects with clinically significant changes in Electrocardiogram (ECG)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Leona P Mörschel, Principal Investigator — Profil Mainz GmbH
Locations (1):
- Profil Mainz GmbH, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No